CLINICAL TRIAL: NCT05473767
Title: Expanding the Family Check-Up in Early Childhood to Promote Cardiovascular Health of Mothers and Young Children (ENRICH)
Brief Title: Expanding the Family Check-Up in Early Childhood to Promote Cardiovascular Health of Mothers and Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Janet Catov, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY22020096; 1UG3HL163116-01 (NIH)
Record Dates: First submitted 2022-07-19; First posted 2022-07-26 (Actual); Results first posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-11

CONDITIONS: Obesity, Maternal; Hypertension in Pregnancy; Hypertension, Pregnancy-Induced; Diabetes; Overweight
Keywords: Cardiovascular health; Postpartum women; Health Promotion
MeSH Terms: conditions — Pregnancy in Obesity; Hypertension, Pregnancy-Induced; Diabetes Mellitus; Overweight

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial pilot study that will randomize 100 women into Family Check-Up Heart and 50 women into traditional Family Check-Up. The investigators will use an unbalanced design to enhance ability to evaluate feasibility and acceptability for the new Family Check-Up Heart intervention. The investigators will utilize a Type 1 hybrid effectiveness-implementation design using mixed methods that will simultaneously assess both the implementation of the Family Check-Up Heart and preliminary effectiveness on 6-month maternal cardiovascular health outcomes.
Who Masked: Investigator
Masking Description: Investigators will be blind to group assignment during intervention delivery and assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Check Up Control (Active Comparator): The Family Check-Up is a home visiting program that typically takes place over the course of 3-5 sessions - An initial interview, assessment, feedback session, and optional treatment sessions. The Family Check-Up is designed to support child development and improve parental well-being.
  Interventions: Behavioral: Family Check-Up
- Family Check-Up Heart (Experimental): Family Check-Up Heart combines the traditional Family Check-Up with a heart health component.
  Interventions: Behavioral: Family Check Up Heart

INTERVENTIONS:
Behavioral: Family Check Up Heart — Family Check-Up Heart consists of the Family Check up with an added heart health component. The Family Check-Up Heart assessment will include evaluations of maternal cardiovascular health; specifically, measurement of maternal blood pressure, body mass index, diet quality, exercise, and smoking, which will be included in the feedback session. After the Feedback Session participants will also receive information about healthy eating and weight loss, stress management, and smoking and to monitor weight and blood pressure.
  Arms: Family Check-Up Heart
Behavioral: Family Check-Up — The Family Check-Up typically takes place over the course of 3-5 sessions, each about an hour long. First, a trained Family Check-Up family coach will conduct an "Initial Interview." Second is an assessment of that includes questionnaires and videotaped interaction tasks. Third, during the Feedback Session, the family coach discusses with the participant strengths and challenges for their child and family as a whole. They then set goals for their family to support and maintain strengths, and to address any areas of concern. After the Feedback Session families have the option to continue meeting with their family coach to support the child's development and improve parental well-being.
  Arms: Family Check Up Control

SUMMARY:
This randomized-controlled pilot study will examine the implementation of a cardiovascular health intervention on postpartum mothers and infants. The investigators will adapt a cardiovascular health intervention into an evidence-based home visiting program, Family Check-Up to create Family Check-Up Heart. Through a Type 1 hybrid effectiveness implementation design, the pilot study will test the feasibility and effectiveness of Family Check-Up Heart (Family Check-Up Heart, n=100; Family Check-Up, n=50). The investigators hypothesize that Family Check-Up Heart will show comparable levels of engagement and acceptability as Family Check-Up alone, and mothers receiving Family Check-Up Heart will have greater improvements in cardiovascular health at 6 months postpartum compared to Family Check-Up alone.

DETAILED DESCRIPTION:
This randomized-controlled pilot study will examine the implementation of a cardiovascular health intervention on pregnant and postpartum mothers. The investigators will adapt a cardiovascular health intervention into an evidence-based home visiting program, Family Check-Up to create Family Check-Up Heart. Through a Type 1 hybrid effectiveness implementation design, the pilot study will test the feasibility and effectiveness of Family Check-Up Heart (Family Check-Up Heart, n=100; Family Check-Up, n=50). The investigators hypothesize that Family Check-Up Heart will show comparable levels of engagement and acceptability as Family Check-Up alone, and mothers receiving Family Check-Up Heart will have greater improvements in cardiovascular health at 6 months postpartum compared to Family Check-Up alone.

A second goal of the hybrid study is to understand the reach, engagement, and context for implementation of Family Check-Up Heart and gather information for development of the multi-center home visiting model trial. The Family Check-Up Heart program is intended to improve the cardiovascular health of low-income mothers compared to the traditional Family Check-Up and other home visiting programs by incorporating individualized, culturally competent interventions that target diet and exercise, blood pressure control, stress management and self-care, and smoking cessation. The intervention includes cardiovascular assessment and feedback, followed by a tailored treatment program delivered by family coaches in 3-4 week modules to establish goals and track progress. These sessions will work towards obtaining positive cardiovascular health outcomes and empowering mothers of infants to achieve their goals through education and a connection to resources which the investigators hypothesize will also preserve child cardiovascular health. Primary analyses will assess the impact of Family Check-Up Heart on maternal cardiovascular health outcomes when the child is 6 months old compared to Family Check-Up alone.

ELIGIBILITY:
Inclusion Criteria:

* Adult inclusion criteria:

  1. Pregnant women/birthing people or women/birthing people who have delivered in the past 2 months who deliver at Magee or are enrolled in the Women Infants and Children program in Allegheny County.
  2. Medicaid-eligible
  3. Speak English.
  4. Resident of Allegheny County, Pennsylvania.
  5. Does not have complex, on-going conditions such as chronic renal or liver disease, systemic lupus erythematosus, cancer or HIV.

Participants who consent to enrollment may have their medical history reviewed by study physicians and staff to adjudicate pregnancy outcomes and ensure they meet inclusion criteria before randomization.

Child inclusion criteria:

1. Children birth through 2 months who reside in Allegheny County may enroll in the program if their mother is participating in the study.
2. Has a legal guardian who speaks English. This criterion is included because the project's materials and assessments are currently only available in English, with staff only fluent in English.

Exclusion Criteria:

1. Pregnant women with complex, on-going conditions such as chronic renal or liver disease, systemic lupus erythematosus, cancer or HIV.
2. Multifetal pregnancies or deliveries.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet M Catov, PhD, Principal Investigator — UPMC Magee Womens Hospital
Locations (3):
- United States (3):
  - Healthy Start, Inc., Pittsburgh, Pennsylvania
  - Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Women, Infants, and Children Program, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Following the requirements of the University of Pittsburgh Institutional Review Board, investigators may access de-identified data following request and approval by the study Principle Investigators. All data will be shared, except when deemed protected health information. For example, maternal age at delivery will be shared by not date of birth or date of delivery (only year). The Principle Investigators will oversee data sharing to ensure no personally identifiable information is shared, and the study data manager has protocols to implement these processes.
Time Frame: We will share data within two years of the end of our funding to allow time for analysis and dissemination of findings.
Access Criteria: Interested investigators seek written approval from the study Principle Investigators. An Institutional Review Board protocol approved by their institution or a signed data sharing agreement is needed to access the data.

REFERENCES:
- [Background] Segal-Isaacson CJ, Wylie-Rosett J, Gans KM. Validation of a short dietary assessment questionnaire: the Rapid Eating and Activity Assessment for Participants short version (REAP-S). Diabetes Educ. 2004 Sep-Oct;30(5):774, 776, 778 passim. doi: 10.1177/014572170403000512. No abstract available. PMID 15510530
- [Background] Chasan-Taber L, Schmidt MD, Roberts DE, Hosmer D, Markenson G, Freedson PS. Development and validation of a Pregnancy Physical Activity Questionnaire. Med Sci Sports Exerc. 2004 Oct;36(10):1750-60. doi: 10.1249/01.mss.0000142303.49306.0d. PMID 15595297

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In person and remote recruitment at several locations serving pregnant women and mothers with newborns including a large birthing hospital and WIC clinics. Eligibility criteria: (1) Single pregnancy or biological mother of child < 2 months old, (2) Allegheny County, PA residency, (3) Medicaid or WIC receipt, (4) English fluency, (5) is/will be main caretaker of the baby in their home, and (6) no complex medical conditions. Participants were randomized 2:1 to the intervention after consent.
Period: Overall Study
Arm/Group | Family Check Up Control | Family Check-Up Heart
Started | 30 | 87
Completed | 15 | 54
Not Completed | 15 | 33

BASELINE CHARACTERISTICS:
Population: 23 participants enrolled in the study but did not complete baseline questionnaires.
Groups:
- Total: Total of all reporting groups
Arm/Group | Family Check Up Control | Family Check-Up Heart | Total
Number analyzed (Participants) | 23 | 71 | 94
Age, Continuous [Mean (Standard Deviation); unit: Year] — Age at enrollment was calculated using participant's date of birth.
  Year | 28.3 (6.85) | 29.7 (5.20) | 29.4 (5.64)
Sex: Female, Male [Count of Participants; unit: Participants] — Parent self-report.
  Participants
    Female | 23 | 71 | 94
    Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Parent self-report. What do you identify as your race(s)? Please select ALL that apply.
  Participants
    American Indian or Alaska Native | 2 | 2 | 4
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 13 | 39 | 52
    White | 7 | 22 | 29
    More than one race | 1 | 8 | 9
    Unknown or Not Reported | 0 | 0 | 0
Weight at 4 weeks postpartum [Mean (Standard Deviation); unit: Pounds] — Weight at 4 weeks postpartum assessed using validated Bluetooth devices Population: Fewer participants were assessed for in person weight measurements.
  Pounds
    number analyzed (Participants) | 20 | 52 | 72
    (all) | 186.43 (63.79) | 200.53 (56.30) | 196.76 (58.27)
Pre-pregnancy weight [Mean (Standard Deviation); unit: Pounds] — Assessed as part of a pregnancy history assessment. "What was your pre-pregnancy weight (in pounds)?" Population: Fewer participants were assessed for the staff-led interview.
  Pounds
    number analyzed (Participants) | 20 | 59 | 79
    (all) | 181.7 (63.5) | 200.6 (60.5) | 196.6 (61.0)
Blood pressure (Systolic) at 4 weeks postpartum assessed using validated Bluetooth devices [Mean (Standard Deviation); unit: Systolic mmHg] — Population: Fewer participants were assessed for in person blood pressure measurements.
  Systolic mmHg
    number analyzed (Participants) | 19 | 52 | 71
    (all) | 115.05 (17.97) | 120.92 (14.30) | 119.35 (15.45)
Blood pressure (Diastolic) at 4 weeks postpartum assessed using validated Bluetooth devices [Mean (Standard Deviation); unit: Diastolic mmHg] — Population: Fewer participants were assessed for in person blood pressure measurements.
  Diastolic mmHg
    number analyzed (Participants) | 19 | 52 | 71
    (all) | 77.84 (10.38) | 83.79 (12.21) | 82.20 (11.97)
BMI at 4 weeks postpartum [Mean (Standard Deviation); unit: kg/m^2] — Weight was assessed using a validated Bluetooth scale and height was assessed via parent report - How tall are you in feet and inches? Population: Fewer participants were assessed for in person weight measurements.
  kg/m^2
    number analyzed (Participants) | 20 | 52 | 72
    (all) | 29.5 (12.46) | 32.73 (8.97) | 31.83 (10.10)
Rapid Eating Assessment for Participants (REAP) - Shortened Version [Mean (Standard Deviation); unit: Score (13-39)] — The REAP is a 16-item self-report scale assessing frequency of various eating behaviors such as skipping breakfast and eating fried foods. Items are rated on a 3-point response scale ranging from Usually/Often (1) to Rarely/Never (3). Three items also have a "Does not apply to me" option which is coded as a 3. The first 13 items are summed to create a score where higher values indicate healthier eating behaviors. Minimum and maximum scores are 13 and 39, respectively. Population: Two participants in the FCU Heart group did not complete the questionnaire.
  Score (13-39)
    number analyzed (Participants) | 23 | 69 | 92
    (all) | 27.43 (3.46) | 26.9 (3.59) | 27.10 (3.54)
Pregnancy Physical Activity Questionnaire (PPAQ) [Mean (Standard Deviation); unit: Score (0-308.85)] — The PPAQ is a 26-item self-report of activities such as jogging, dancing, and watching television. Items are rated on a 6-point likert-type scale (Never to 3 or more hours/day). Responses are weighted, generating metabolic equivalent codes (time spent in each activity is multiplied by its intensity to derive average weekly energy expenditure for each activity). The metabolic equivalent codes are summed to create a physical activity score where higher values indicate greater activity. Minimum and maximum scores are 0 and 308.85, respectively.
  Score (0-308.85) | 89.45 (65.91) | 101.55 (59.72) | 98.52 (61.19)

OUTCOME MEASURES:

1. Primary Outcome: Change in Postpartum Weight Retention
Description: Weight change from post-delivery to 6 months; both will be measured by the study using validated Bluetooth devices and following standardized research protocols. Mean difference scores are reported.
Time Frame: Baseline to 6 months post-partum
Population: Participants who were retained for outcomes assessment were used in analyses.
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | Family Check Up Control | Family Check-Up Heart
Number analyzed (Participants) | 13 | 46
Pounds | -.73 (9.9) | .29 (14.1)

2. Secondary Outcome: Weight at 6 Months Postpartum
Description: Weight at 6 months will be assessed by the study using validated Bluetooth devices and following standardized research protocols.
Time Frame: 6 months post-partum
Population: Participants who were retained for outcomes assessment were used in analyses.
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | Family Check Up Control | Family Check-Up Heart
Number analyzed (Participants) | 13 | 46
Pounds | 200.2 (70.9) | 202.1 (58.3)

3. Secondary Outcome: Weight Change From First Measured Prenatal Weight to 6 Months Postpartum
Description: First measured prenatal weight will be obtained from the participant's medical record at baseline. Weight at 6 months will be assessed by the study using validated Bluetooth devices and following standardized research protocols. Mean difference scores are reported.
Time Frame: Baseline to 6 months post-partum
Population: Participants who were retained for outcomes assessment were used in analyses.
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | Family Check Up Control | Family Check-Up Heart
Number analyzed (Participants) | 13 | 46
Pounds | 11.5 (15.2) | 1.98 (18.9)

4. Secondary Outcome: Change in Self-reported Pre-pregnancy Weight to 6 Months Postpartum
Description: Pre-pregnancy weight will be self-reported at the baseline assessment. Weight at 6 months post-partum will be assessed by the study using validated Bluetooth devices and following standardized research protocols. Mean difference scores are reported.
Time Frame: Baseline to 6 months post-partum
Population: Participants who were retained for outcomes assessment were used in analyses.
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | Family Check Up Control | Family Check-Up Heart
Number analyzed (Participants) | 13 | 46
Pounds | 13.1 (24.2) | 4.7 (24.2)

5. Secondary Outcome: Change in Blood Pressure From Post-delivery to 6 Months.
Description: Blood pressure will be measured by the study at baseline and again at 6-months post-partum using validated Bluetooth devices and following standardized research protocols. Mean difference scores are reported.
Time Frame: Baseline to 6 months post-partum
Population: Participants who were retained for outcomes assessment were used in analyses.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Family Check Up Control | Family Check-Up Heart
Number analyzed (Participants) | 13 | 46
mmHg
  Systolic mmHg | -1.76 (7.4) | -1.4 (13.5)
  Diastolic mmHg | -1.38 (6.8) | -3.59 (13.2)

6. Secondary Outcome: Change in Blood Pressure From First Prenatal Visit to 6 Months.
Description: First measured prenatal blood pressure will be obtained from the participant's medical record at baseline. Blood pressure at 6 months post-partum will be assessed by the study using validated Bluetooth devices and following standardized research protocols. Mean difference scores are reported.
Time Frame: Baseline to 6 months post-partum
Population: Participants who were retained for outcomes assessment were used in analyses.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Family Check Up Control | Family Check-Up Heart
Number analyzed (Participants) | 13 | 46
mmHg
  Systolic mmHg | -6.3 (12.8) | -.20 (14.4)
  Diastolic mmHg | 8.3 (12.2) | 8.8 (11.7)

7. Secondary Outcome: Blood Pressure at 6 Months Post-partum
Description: Blood pressure at 6 months post-partum will be assessed by the study using validated Bluetooth devices and following standardized research protocols.
Time Frame: 6 months post-partum
Population: Participants who were retained for outcomes assessment were used in analyses.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Family Check Up Control | Family Check-Up Heart
Number analyzed (Participants) | 13 | 46
mmHg
  Systolic mmHg | 117.4 (15.4) | 119.1 (12.5)
  Diastolic mmHg | 78.5 (11.4) | 79.8 (9.0)

8. Secondary Outcome: BMI at 6 Months Post-partum
Description: Height and Weight at 6 months post-partum will be assessed by the study using a validated Bluetooth scale and following standardized research protocols.
Time Frame: 6 months post-partum
Population: Participants who were retained for outcomes assessment were used in analyses.
Measure: Mean (Standard Deviation); unit: kg/m²
Arm/Group | Family Check Up Control | Family Check-Up Heart
Number analyzed (Participants) | 13 | 46
kg/m² | 32.7 (12.5) | 32.9 (9.2)

9. Secondary Outcome: Change in Eating Behaviors
Description: Eating behaviors will be assessed at baseline and 6 months post-partum using the Rapid Eating Assessment for Participants - Shortened Version. The Rapid Eating Assessment for Participants is a 16-item self-report scale assessing frequency of various eating behaviors such as skipping breakfast and eating fried foods. Items are rated on a 3-point response scale ranging from Usually/Often (1) to Rarely/Never (3). Three items also have a "Does not apply to me" option which is also coded as a 3. An example of an item with this option is "Eat more than 8 ounces of meat, chicken, turkey, or fish per day." The first 13 items are summed to create a score where higher values indicate healthier eating behaviors. Minimum and maximum scores are 13 and 39, respectively. Mean difference scores are reported.
Time Frame: Baseline to 6 months post-partum
Population: Participants who were retained for outcomes assessment were used in analyses.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Family Check Up Control | Family Check-Up Heart
Number analyzed (Participants) | 13 | 46
Score | -.50 (4.1) | .39 (3.8)

10. Secondary Outcome: Change in Physical Activity
Description: Physical activity will be measured using the Pregnancy Physical Activity Questionnaire. The Pregnancy Physical Activity Questionnaire is a 26-item self-report of activities such as jogging or running, dancing, and watching television or a video. Items are rated on a 6-point likert-type scale ranging from Never to 3 or more hours per day. Responses are weighted to generate metabolic equivalent codes. Specifically, the self-reported time spent in each activity will be multiplied by its intensity to arrive at a measure of average weekly energy expenditure attributable to each activity. The metabolic equivalent codes are then summed to create a physical activity score where higher values indicate greater physical activity. Minimum and maximum scores are 0 and 308.85, respectively. Mean difference scores are reported.
Time Frame: Baseline to 6 months post-partum
Population: Participants who were retained for outcomes assessment were used in analyses.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Family Check Up Control | Family Check-Up Heart
Number analyzed (Participants) | 13 | 46
Score | 20.2 (91.1) | 27.8 (75.8)

ADVERSE EVENTS:
Time Frame: AE assessment occurred at all intervention sessions.
Description: Adverse events were monitored from enrollment to 6 months postpartum via clinical check-ins at each intervention session. Sessions included an initial interview, monthly phone check-ins during pregnancy, a feedback session, and optional monthly sessions until study end. Caregivers were asked whether they experienced any emotional/psychological or physical difficulties related to study participation. Research staff also monitored for distress at the 6-month assessment.
Arm/Group | Family Check Up Control | Family Check-Up Heart
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/87
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/87
Other Adverse Events (participants affected / at risk) | 0/30 | 0/87

LIMITATIONS AND CAVEATS:
Limitations of the study include the small sample size and the short duration of intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/67/NCT05473767/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/67/NCT05473767/SAP_001.pdf
  • Informed Consent Form (2023-07-07): https://cdn.clinicaltrials.gov/large-docs/67/NCT05473767/ICF_002.pdf